CLINICAL TRIAL: NCT03593278
Title: Single-center, Open-label Study With 14C-radiolabeled ACT-246475 to Investigate Its Mass Balance, Pharmacokinetics, and Metabolism Following Single Subcutaneous Administration to Healthy Male Subjects
Brief Title: A Study to Evaluate ACT-246475 Fate in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ID-076-104; 2017-004622-15 (EudraCT Number)
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2022-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — selatogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment and observation period (Experimental): On Day 1, the subjects will receive a single s.c. dose of 16 mg 14C-radiolabeled ACT-246475 in the fasted state. Subjects will be followed by an observation period of 3 days (72 h) during which blood, urine, and feces samples will be collected.
  Interventions: Drug: ACT-246475

INTERVENTIONS:
Drug: ACT-246475 — Single s.c. dose of 16 mg ACT-246475 including 3.7 MBq (100 μCi) 14C-radiolabeled ACT 246475

SUMMARY:
The purpose of this study is to investigate how quickly and to what extent ACT-246475 is absorbed, distributed, metabolized (broken down) and eliminated from the body. ACT-246475 will be labeled with 14-Carbon (14C) and, in this way can be traced in blood, urine, and feces. This study will also investigate how safe is ACT-246475 and how well it is tolerated when administered to healthy male volunteers.

ELIGIBILITY:
Main Inclusion Criteria:

* Signed informed consent in the local language prior to any studymandated procedure,
* Healthy male subjects aged between 45 and 65 years (inclusive) at screening,
* No clinically significant findings on the physical examination at screening,
* Body mass index of 18.0-28.0 kg/m2 (inclusive) at screening,
* Systolic blood pressure (BP) 100-140 mmHg, diastolic BP 50-90 mmHg, and pulse rate 45-90 bpm (inclusive), measured on either arm, after 5 min in the supine position at screening,
* 12-lead electrocardiogram (ECG) without clinically relevant abnormalities, measured after 5 min in the supine position at screening,
* Values of closure time tested with the Platelet Function Analyzer equipment, for both cartridges of collagen/epinephrine and collagen/adenosine diphosphate below the upper limit of normal range at screening.

Main Exclusion Criteria:

* Known hypersensitivity to ACT-246475 or drugs of the same class, or any excipients of the ACT-246475 formulation,
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study treatment (appendectomy and herniotomy allowed, cholecystectomy not allowed),
* Family or personal history of prolonged bleeding (e.g., after surgical intervention) or bleeding disorders (e.g., thrombocytopenia, clotting disturbances), intracranial vascular diseases, stroke, reasonable suspicion of vascular malformations, or peptic ulcers,
* Platelet count < 120 x10^9 L-1 at screening,
* Previous exposure to ACT-246475,
* Participation in another study with a radiation burden of > 0.1 mSv and ≤ 1.0 mSv in a period of 1 year prior to screening; a radiation burden of > 1 mSv and ≤ 2.0 mSv in a period of 2 years prior to screening, etc. (add 1 year per 1 mSv),
* Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton [excluding spinal column]), during work or during participation in a clinical study, in the period of 1 year prior to screening,
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2018-08-05 (Actual); Study Completion 2018-08-05 (Actual)

PRIMARY OUTCOMES:
Cumulative excretion of total 14C-radioactivity in urine and feces | Up to 54 days
  Cumulative amount of total 14C-radioactivity excreted in urine and feces will be calculated by summing up the amount of total 14C-radioactivity of the samples excreted in each collection interval

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (3):
- Germany (3):
  - Universitäts-Herzzentrum Bad Krozingen, Bad Krozingen
  - Universitäts-Herzzentrum Freiburg, Freiburg im Breisgau
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen

IPD SHARING:
Plan to Share IPD: No